CLINICAL TRIAL: NCT03427424
Title: Imaging Biomarker for Addiction Treatment Outcome
Status: Terminated | Type: Observational
Why Stopped: Lab staffing changes and the COVID pandemic affected resources in such a way that the study could not be completed.
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999918053; 18-DA-N053
Record Dates: First submitted 2018-02-08; First posted 2018-02-09 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Opioid-Related Disorders; Alcohol-Related Disorders
Keywords: Opioid use Disorder; Alcohol Use Disorder; Physician Health Program; Functional Magnetic Resonance Imaging (fMRI); Magnetic Resonance Spectroscopy; Natural History
MeSH Terms: conditions — Opioid-Related Disorders; Alcohol-Related Disorders; Alcoholism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (8):
- AUD-E: Early-in-treatment, healthy alcohol use disorder participants currently enrolled in PHP within 2 months of starting treatment (AUD-E)
- AUD-L: Long-term-in-treatment, healthy alcohol use disorder participants currently enrolled in PHP more than 2 months and less than 5 years (AUD-L)
- Characterization: substance use disorder participants currently enrolled in PHP, not eligible for main imaging study
- CON: healthy, non-drug using control participants (CON)
- POAUD-E: Early-in-treatment, healthy dual prescription opioid and alcohol and use disorder participants currently enrolled in PHP within 2 months of starting treatment (POAUD-E)
- POAUD-L: Long-term-in-treatment, healthy dual prescription opioid and alcohol use disorder participants currently enrolled in PHP more than 2 months and less than 5 years (POAUD-L)
- POUD-E: Early-in-treatment, healthy prescription opioid use disorder participants currently enrolled in physician health program (PHP) within 2 months of starting treatment (POUD-E)
- POUD-L: Long-term-in-treatment, healthy prescription opioid use disorder participants currently enrolled in PHP more than 2 months and less than 5 years (POUD-L)

SUMMARY:
Background:

Many people suffer from drug addiction. But currently, treatments are not very effective. One group of patients in this study are enrolled in addiction treatment through physician health programs (PHPs). About 70% of these patients are able to stop using drugs for extended periods of time. By studying this specific group of patients, researchers want to understand the difference between those who may or may not respond to treatment. They want to study the brain while people do thinking and feeling tasks and when they relax. They will study brain chemicals, a stress hormone, and certain genes. The results may help them understand the brain basis for addiction and recovery.

Objectives:

To use brain imaging to find differences between people with and without drug addiction. To see if these differences help predict addiction.

Eligibility:

Healthy, right-handed adults ages 21-65, enrolled in a physician health program or those with no history of addiction and with at least 16 years of education

Design:

Participants enrolled in a PHP will be screened under this study and participants with no history of addiction will be screened under another study.

At the study visit, participants will:

Have a routine check-up, including tests for pregnancy, drugs, and alcohol.

Give 11 blood samples.

Rate their cravings.

Test their frustration with stressful situations by responding to questions on a screen.

Practice the magnetic resonance imaging (MRI) tasks:

Shock task. Two electrodes placed on a foot will deliver brief, low-strength electrical shocks that get gradually stronger, but not painful. Participants will see drug or neutral images. They will rate their discomfort.

Thinking tasks. Participants will answer questions about pictures, numbers, and money. They will press buttons in response to things they see.

Do the MRI tasks in 2 sessions (morning and afternoon) in the scanner. Participants will lie in an MRI machine which will take pictures of the brain while doing these tasks.

Some participants will repeat the visit twice over a year at set intervals.

Meals will be provided, and visits will include meal breaks and smoking breaks for those who smoke.

DETAILED DESCRIPTION:
Objective:

Despite recent advances in addiction neuroscience, achieving a breakthrough in predicting addiction treatment outcome has been difficult and long-term abstinence success unacceptably low. The aim of this study is to create a biomarker using various neuroimaging metrics that can predict treatment outcome in opioid, alcohol and dual opioid and alcohol use disorder patients.

Study Population:

Total study enrollment will include up to 650 participants. The main study population will include up to five hundred (500) participants to reach three hundred fifty (350) completers (50 per group) based on their addiction status (1) healthy, non-drug using control participants (CON) (2) Early-in-treatment, healthy prescription opioid use disorder participants currently enrolled in physician health program (PHP) within 3 months of starting treatment (POUD-E), (3) Long-term-in-treatment, healthy prescription opioid use disorder participants currently enrolled in or affiliated with a PHP more than 2 months (POUD-L), (4) Early-in-treatment, healthy alcohol use disorder participants currently enrolled in PHP within 3 months of starting treatment (AUD-E), (5) Long-term-in-treatment, healthy alcohol use disorder participants currently enrolled in or affiliated with a PHP more than 2 months (AUD-L), (6) Early-in-treatment, healthy dual prescription opioid and alcohol and use disorder participants currently enrolled in PHP within 3 months of starting treatment (POAUD-E), (7) Long-term-in-treatment, healthy dual prescription opioid and alcohol use disorder participants currently enrolled in or affiliated with a PHP more than 2 months (POAUD-L). The Addiction Phenotype Characterization arm will include up to 150 completers.

Design:

The main study includes two studies that will run simultaneously:

Cross-sectional study that will include participants who have been in treatment for more than 2 months and are either enrolled at a PHP if within the required monitoring period of 5 years or still affiliated with their PHP after successfully completing their 5-year monitoring period. Three target groups, in addition to the control group, will be included in this study [POUD-L, AUD-L, and POAUD-L]. Each participant will complete a screening evaluation session (approximately 3-4 hours) and a second session for study consent review (approximately 1-2 hours) at home or at the PHP through secure communication. These sessions will include the screening consent process, administration of a structured psychiatric interview and a semi-structured assessment, instructions for the completion of detailed self-administered questionnaires to characterize clinical phenotype and physical condition, and consent review for the study. Participants subsequently cleared for and enrolled in the cross-sectional study will be invited to come to NIDA IRP for one imaging visit that will take approximately 8-10 hours.

The aim of the cross-sectional study is to identify imaging based brain differences between control group and drug using groups and to examine correlations between brain imaging markers at different stages of recovery and (1) severity of drug use (duration and quantity), (2) duration of abstinence, and (3) number of relapses in drug using groups.

The primary outcome measure for the cross-sectional study will be differences in functional connectivity and BOLD signal activation in executive and impulsive neurobehavioral decision systems at various stages of sobriety in relation to controls.

Longitudinal study that will include participants who are enrolled at a PHP within about three months of starting treatment. Three groups, in addition to the control group, will be included in this study [POUD-E, AUD-E, and POAUD-E]. Each participant will complete the screening sessions as described in the cross-sectional study. Eligible participants will undergo three imaging visits at NIDA; 1) 1st (baseline) visit within about 2 months of eligibility determination, (2) 2nd (mid-year) visit within 4-8 months of baseline visit and (3) 3rd (one-year) visit within 10-14 months of baseline visit. Each imaging visit will take approximately 8-10 hours.

The aim of the longitudinal study is to measure brain imaging changes over time in abstinent and relapsing addicts and to identify brain imaging markers that differentiate between abstinent and relapsing participants at 6 months and at 1 year. The rationale behind the mid-year visit is that most relapses take place early (within the first 6 months) during treatment and, by one year, some of those who relapsed earlier achieve abstinence. We chose one year follow up in order to compare brain imaging changes between abstinent and relapsing participants after relatively long sobriety and to add clinical value to our prediction model. By including both of these visits, we will obtain three scans on both abstinent without early relapse and abstinent with early relapse in order to uncover salient brain differences between those who relapse early and those who maintain abstinence.

The primary outcome measure for the longitudinal study will be differences in baseline and changes over time in functional connectivity circuits and BOLD signal activation in executive and impulsive neurobehavioral decision systems between abstinent and relapsing addicts that can predict treatment response at 6 and 12 months. Most importantly, we will use imaging, behavioral and genetic measures at the onset of treatment in a machine-learning framework in an attempt to predict subsequent treatment success in this cohort of participants.

Secondary outcome measures for both studies will be phenotypic (performance on behavioral tasks, self-reported measures of cravings, impulsivity and personality traits), genotypic and imaging (structural, functional and spectroscopy) differences between different addiction groups.

The Addiction Phenotype Characterization arm will include participants who are ineligible for the main study due to imaging-related exclusions or other medical exclusions (e.g. medications, other SUD disorders). These participants will complete the characterization measures (structured psychiatric interview, a semi-structured drug use history assessment, and several self-administered questionnaires to characterize clinical phenotype and physical condition).

The aim of the Addiction Phenotype Characterization arm is to characterize addiction phenotype and physical condition in health professionals.

The primary outcome measures for the Addiction Phenotype Characterization arm are the characterization measures.

ELIGIBILITY:
* I. MAIN STUDY

A. INCLUSION CRITERIA:

All participants: (CON), (POUD-E), (POUD-L), (AUD-E), (AUD-L), (POAUD-E), (POAUD-L):

* Males and females between 21-65 years of age will be enrolled in the study.
* Able and willing to provide written informed consent.
* Must be right-handed.
* Participants must be in good health.

Healthy control participants (CON) in addition to all participants inclusion criteria:

* Free of lifetime DSM-5 substance use disorders except for tobacco use disorder.
* 16 years of education or more

Early-in-treatment, prescription opioid use disorder (POUD-E) participants- in addition to all participants inclusion criteria:

* Recently (within about 3 months) enrolled in a physician health program (PHP) or equivalent at time of enrollment in the study.
* Meet a minimum of 6/11 DSM-5 criteria for severe opioid use disorder (OUD) for about 2 years prior to enrollment and abstinent for about 1-3 months at time of imaging.

Early-in-treatment, alcohol use disorder (AUD-E) participants- in addition to all participants inclusion criteria

* Recently (within about 3 months) enrolled in a physician health program (PHP) or equivalent at time of enrollment in the study.
* Meet a minimum of 6/11 DSM-5 criteria for severe alcohol use disorder (AUD) for about 2 years prior to enrollment and abstinent for about 1-3 months at time of imaging.

Early-in-treatment, dual prescription opioid and alcohol use disorder (POAUD-E) participants- in addition to all participants inclusion criteria:

* Recently (within about 3 months) enrolled in a physician health program (PHP) or equivalent at time of enrollment in the study.
* Meet a minimum of 6/11 DSM-5 criteria for either severe opioid or severe alcohol use disorders and a minimum of 4/11 DSM-5 for either moderate opioid or moderate alcohol use disorder for about 2 years for each substance prior to enrollment and abstinent for about 1-3 months at time of imaging.

Long-term-in-treatment, prescription opioid use disorder (POUD-L) participants- in addition to all participants inclusion criteria:

* Enrolled in or affiliated with a physician health program (PHP) or equivalent for more than 2 months at time of enrollment in the study.
* Meet a minimum of 6/11 DSM-5 criteria for severe opioid use disorder for about 2 years prior to starting treatment and abstinent for at least 3 months at time of imaging.

Long-term-in-treatment, alcohol use disorder (AUD-L) participants- in addition to all participants inclusion criteria:

* Enrolled in or affiliated with a physician health program (PHP) or equivalent for more than 2 months at time of enrollment in the study and in full remission for at least 2 months at time of imaging.
* Meet a minimum of 6/11 DSM-5 criteria for severe alcohol use disorder for about 2 years prior to starting treatment and abstinent for at least 3 months at time of imaging.

Long-term-in-treatment, dual prescription opioid and alcohol use disorder (POAUD-L) participants - in addition to all participants inclusion criteria:

* Enrolled in or affiliated with a physician health program (PHP) or equivalent for more than 2 months at time of enrollment in the study.
* Meet a minimum of 6/11 DSM-5 criteria for either severe opioid or severe alcohol use disorder and a minimum of 4/11 DSM-5 for either moderate opioid or moderate alcohol use disorder about 2 years for each substance prior to enrollment and abstinent for at least 3 months at time of imaging.

EXCLUSION CRITERIA:

All participants: (CON), (POUD-E), (POUD-L), (AUD-E), (AUD-L), (POAUD-E), (POAUD-L):

* Females must not be pregnant or lactating.
* Presence of ferromagnetic objects in the body that are contraindicated for MRI of the head (e.g. pacemakers or other implanted electrical devices, brain stimulators, some types of dental implants, aneurysm clips, metallic prostheses, permanent eyeliner, implanted delivery pump, or shrapnel fragments) or fear of enclosed spaces.
* Noise-induced hearing loss or tinnitus.
* Head trauma with loss of consciousness for more than 30 minutes or significant sequelae for more than one month.
* Current or past DSM-5 diagnosis of any psychiatric disorder that required hospitalization other than detoxification (any length), or chronic medication management for more than three months, (except for stable doses of antidepressants, or low dose (up to 100mg/day of Quetiapine or equivalent) of antipsychotics (experimental groups only) for at least one month prior to the time of a scanning visit) and that could impact brain function at the time of the study based on study MAI s discretion. Current or past tobacco use disorder or nicotine use, opioid use disorder in opioid use disorder participants, alcohol use disorder in alcohol use disorder participants, and both opioid and alcohol use disorders in the dual opioid and alcohol use disorder group is not exclusionary.
* Currently (at time of imaging sessions) using any medications that are known to alter BOLD signal such as stimulant or stimulant-like medications (amphetamine, methylphenidate, modafinil); anorexics (sibuteramine); antianginal agents; antiarrhythmics; antiasthma agents that are systemic corticosteroids; anticholinergics; anticonvulsants; antineoplastics; antiobesity; hormones (exceptions: thyroid hormone replacement, oral contraceptives, and estrogen replacement therapy); insulin; lithium; herbal products with known psychotropic effects (e.g. Gingko biloba, or St. John s Wort) and other medications based on study MAI s discretion.
* Currently (at time of imaging sessions) taking methadone opioid replacement therapy. Please note that experimental group participants taking disulfiram, acamprosate, naltrexone, or long acting naltrexone treatment or those at a stable dose (for at least 2 weeks) of buprenorphine containing medications will be allowed to participate in the study.
* Medical conditions that can impact brain function such as seizure disorder, diabetes mellitus, renal insufficiency (e.g. Creatinine > 2.5), uncontrolled hypertension (BP> 160/100 on screening), clinically significant heart disease, HIV, syphilis, or autoimmune disorders.
* Clinically significant laboratory results (e.g. random glucose > 200 mg/dL, LFT (ALT, AST and GGT) > 3-fold upper limit of normal, or Hemoglobin < 10 gm/dL) or other clinically significant lab abnormalities based on study MAI s discretion.
* Have any current neurological illnesses including, but not limited to, seizure disorders, frequent migraines or on prophylaxis, multiple sclerosis, movement disorders, or CNS tumor.
* Are non-English speaking.
* Suspected or confirmed acute SARS-CoV-2 infection.

II. ADDICTION PHENOTYPE CHARACTERIZATION

Note: Health professionals with prescription opioid, alcohol or dual prescription opioid and alcohol use disorder or other substances who are enrolled in or affiliated with a PHP and are not eligible for the main study (including for having an SUD that does not qualify for the main study) may be invited to participate in the Addiction Phenotype Characterization arm.

A. INCLUSION CRITERIA:

* Males and females 21 years of age and older will be enrolled in the study.
* Able and willing to provide informed consent.
* Enrolled in or affiliated with a physician health program (PHP) or equivalent at the time of enrollment in the study.
* Meet a minimum of 6/11 DSM-5 criteria for severe opiate, alcohol or both alcohol and opiate or other substance use disorder for at least 2 years prior to enrollment.

B. EXCLUSION CRITERION:

-Are non-English speaking.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Cross-sectional study will include participants enrolled in or affiliated with a PHP for more than 2 months. Longitudinal study will include participants who are enrolled in a PHP within about three months of starting treatment. No preferences in participant recruitment will be made on the bases of gender, race, or ethnic background. Efforts will be made to include minorities in proportion to their presence in the local population of the PHP. The demographic profile for the PHP cohort is about 60% males (Braquehais et al. 2014; Brooks et al. 2013), predominantly Caucasian; 89% and about 4% Asian, 3% Hispanic, 1.5% African American and 1.5% other races (Brooks et al. 2013). The matching control group will be recruited from NIH employees and from the major metropolitan Baltimore area.
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2019-07-10 (Actual); Primary Completion 2024-04-29 (Actual); Study Completion 2024-04-29 (Actual)

PRIMARY OUTCOMES:
For the longitudinal study will be differences in baseline and changes over time in functional connectivity circuits, BOLD signal activation in executive and impulsive neurobehavioral decision systems between abstinent and relapsing addicts that... | 6 & 12 mo f/u visits
  For the longitudinal study will be differences in baseline and changes over time in functional connectivity circuits, BOLD signal activation in executive and impulsive neurobehavioral decision systems between abstinent and relapsing addicts that can predict treatment response at 6 and 12 months.
For the Addiction Phenotype Characterization arm: characterization measures | at completion of characterization measures
  The outcome measures for the Addiction Phenotype Characterization arm are phenotypic factors that are related to addiction as measured by the psychiatric interview, drug use history assessments, and self-administered questionnaires to characterize clinical phenotype and physical condition.
For cross-sectional study will be differences in functional connectivity and BOLD signal activation in executive and impulsive neurobehavioral decision systems at various stages of sobriety in relation to controls | 1 study visit
  For cross-sectional study will be differences in functional connectivity and BOLD signal activation in executive and impulsive neurobehavioral decision systems at various stages of sobriety in relation to controls

SECONDARY OUTCOMES:
Phenotypic (performance on behavioral tasks, self-reported measures of cravings, impulsivity and personality traits), genotypic and imaging (structural and spectroscopy) differences between different addiction groups. | At each visit
  Secondary Outcome Measure: Phenotypic (performance on behavioral tasks, self-reported measures of cravings, impulsivity and personality traits), genotypic and imaging (structural and spectroscopy) differences between different addiction groups.

CONTACTS AND LOCATIONS:
Overall Officials: Amy Janes, Ph.D., Principal Investigator — National Institute on Drug Abuse (NIDA)
Locations (1):
- National Institute on Drug Abuse, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided
.We plan to share IPD for this protocol; however, plans have not yet been finalized. We have not yet finalized decisions on types of supporting information that will be shared, IPD Sharing Time Frame, or IPD Sharing Access Criteria. As stated in the protocol, data will be stripped of identifiers prior to release for sharing. De-identified data may be shared with properly administered databases and/or with collaborators with whom proper data sharing agreements are in place (we will set-up proper data sharing agreements once a plan is determined).